CLINICAL TRIAL: NCT01621048
Title: Evaluation of Treatment Related Toxicity After Radiotherapy for Head and Neck Cancer and Correlation With Dose to Organs at Risk
Brief Title: Evaluation of Treatment Related Toxicity After Radiotherapy for Head and Neck Cancer
Status: Withdrawn | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Sandra Nuyts, Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s54403
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Head and Neck Neoplasms; Xerostomia; Deglutition Disorders
Keywords: Head and Neck Neoplasmsr; Radiotherapy; Xerostomia; Deglutition Disorders
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Radiotherapy plays an important role in the curative treatment of head and neck cancer. This treatment however is associated with significant acute and late toxicity with xerostomia and dysphagia severely implicating the patient's quality of life. With highly conformal radiotherapy techniques it is possible to decrease de dose to the organs at risk while maintaining adequate doses to the tumour. In order to adequately register the effect of these techniques it is imperative to obtain standardized information on the acute and late treatment effects. With this study the investigators want to evaluate this toxicity using standardized and validated questionnaires during follow-up. This data will then be correlated to the doses delivered to the specific organs at risk.

DETAILED DESCRIPTION:
Introduction Radiotherapy is one of the main curative treatment options in advanced head and neck cancer. With the introduction of altered fractionation schedules and concurrent chemotherapy locoregional control numbers and overall survival have improved significantly. This has come at the cost of excess in acute and late toxicity. The steep dose gradients associated with more conformal radiotherapy techniques such as intensity modulated radiotherapy (IMRT) allows us to maintain adequate coverage of the target volume while reducing the dose to the surrounding normal tissues, thus potentially sparing these from excess acute and late toxicity. However to accurately evaluate the value of these new techniques documentation of treatment related toxicity and quality of life is essential. Standardized quality of life scoring systems have been developed for this purpose. Especially xerostomia is very hard to evaluate, although it remains an important issue in the follow-up of these patients.

Purpose In this study the investigators want to analyze treatment related toxicity, with special emphasis on xerostomia and dysphagia in patients treated with radiotherapy for head and neck cancer by presenting them with standardized quality of life questionnaires at well defined points after treatment (2 months, six months, one year ,two years after RT). The result of these questionnaires will then be correlated to treatment data.

Study Design The investigators will include all patient which are in follow-up after primary (chemo-)radiotherapy for head and neck cancer for a period 4 years. At well defined time points after primary (chemo-)radiotherapy for head and neck cancer the investigators will ask the patient to fill in standardized questionnaires compromising of the EORTC QLQ H&N35 questionnaire, the university of Michigan Xerostomia questionnaire (XQ) and the MD Anderson Dysphagia Inventory. The treating physician will score the toxicity using the RTOG/EORTC late toxicity scoring system and the functional oral intake scale (FOIS).

This toxicity data will then be analyzed and correlated with treatment data. Special interest will go to the relationship between the presence of xerostomia and the doses delivered to subvolumes of the parotid glands, the submandibular glands and oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx and larynx.
* Stage T1-4,N0-3; for cancer of the glottis T3-4 or TxN1-3
* Decision for curative radiotherapy or radiochemotherapy made by a multidisciplinary group of head and neck tumors.
* >18 years of age

Exclusion Criteria:

* Previous surgery of the primary tumor or lymph nodes
* Tumour recurrence, locoregional or distant
* Mental condition rendering the patient unable to understand or fill in the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with primary (chemo-)radiotherapy for head and neck squamous cell carcinoma up to 70-72 Gy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
toxicity: EORTC QLQ H&N35 questionnaire, the university of Michigan Xerostomia questionnaire (XQ) and the MD Anderson Dysphagia Inventory. | 5 years
  toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nuyts, M.D., Ph.D, Principal Investigator — Department of Radiotherapy, UZ Gasthuisberg Leuven
Locations (1):
- Department of Radiotherapy-Oncology, UZ Gasthuisberg Leuven, Leuven, Belgium

REFERENCES:
- [Background] Bourhis J, Overgaard J, Audry H, Ang KK, Saunders M, Bernier J, Horiot JC, Le Maitre A, Pajak TF, Poulsen MG, O'Sullivan B, Dobrowsky W, Hliniak A, Skladowski K, Hay JH, Pinto LH, Fallai C, Fu KK, Sylvester R, Pignon JP; Meta-Analysis of Radiotherapy in Carcinomas of Head and neck (MARCH) Collaborative Group. Hyperfractionated or accelerated radiotherapy in head and neck cancer: a meta-analysis. Lancet. 2006 Sep 2;368(9538):843-54. doi: 10.1016/S0140-6736(06)69121-6. PMID 16950362
- [Background] Pignon JP, Bourhis J, Domenge C, Designe L. Chemotherapy added to locoregional treatment for head and neck squamous-cell carcinoma: three meta-analyses of updated individual data. MACH-NC Collaborative Group. Meta-Analysis of Chemotherapy on Head and Neck Cancer. Lancet. 2000 Mar 18;355(9208):949-55. PMID 10768432
- [Background] Nuyts S, Dirix P, Clement PM, Poorten VV, Delaere P, Schoenaers J, Hermans R, Van den Bogaert W. Impact of adding concomitant chemotherapy to hyperfractionated accelerated radiotherapy for advanced head-and-neck squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2009 Mar 15;73(4):1088-95. doi: 10.1016/j.ijrobp.2008.05.042. Epub 2008 Aug 15. PMID 18707823
- [Background] Machtay M, Moughan J, Trotti A, Garden AS, Weber RS, Cooper JS, Forastiere A, Ang KK. Factors associated with severe late toxicity after concurrent chemoradiation for locally advanced head and neck cancer: an RTOG analysis. J Clin Oncol. 2008 Jul 20;26(21):3582-9. doi: 10.1200/JCO.2007.14.8841. Epub 2008 Jun 16. PMID 18559875
- [Background] Nutting CM, Morden JP, Harrington KJ, Urbano TG, Bhide SA, Clark C, Miles EA, Miah AB, Newbold K, Tanay M, Adab F, Jefferies SJ, Scrase C, Yap BK, A'Hern RP, Sydenham MA, Emson M, Hall E; PARSPORT trial management group. Parotid-sparing intensity modulated versus conventional radiotherapy in head and neck cancer (PARSPORT): a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2011 Feb;12(2):127-36. doi: 10.1016/S1470-2045(10)70290-4. Epub 2011 Jan 12. PMID 21236730
- [Background] Dirix P, Nuyts S. Evidence-based organ-sparing radiotherapy in head and neck cancer. Lancet Oncol. 2010 Jan;11(1):85-91. doi: 10.1016/S1470-2045(09)70231-1. PMID 20129131